CLINICAL TRIAL: NCT02454855
Title: Impact of a Melatonin Supplementation on the Quality of Life in Elderly Metastatic Cancer Patients (> = 70 Years) - PHRC-K13-170
Brief Title: Impact of a Melatonin Supplementation on the Quality of Life in Elderly Metastatic Cancer Patients
Acronym: MEQAPAG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study stopped for futility after the DSMB.
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PHRC-K13-170; 2014-003505-14 (EudraCT Number)
Record Dates: First submitted 2015-05-12; First posted 2015-05-27 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: quality of life; melatonin; Elderly patient
MeSH Terms: conditions — Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group "Melatonin" (Experimental): standard anticancer treatment + 3-month of melatonin supplementation
  Interventions: Drug: melatonin
- Group "Placebo" (Placebo Comparator): standard anticancer treatment + placebo (3 months)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: melatonin — Oral supplementation with melatonin (tablets) will be administered for 3 months once daily , 1-2 hours before bedtime. It will start on the day of the first administration of the new line of anticancer treatment (or no later on the day of the second administration of the new line of anticancer treatment).
  Melatonin supplementation is achieved by the administration of (Circadin) at a dose of 2 mg / day according to its MA form of prolonged-release tablet of 2 mg.
  Arms: Group "Melatonin"
Drug: placebo — Oral supplementation with placebo (tablets) will be administered for 3 months once daily , 1-2 hours before bedtime. It will start on the day of the first administration of the new line anticancer treatment (or no later on the day of the second administration of the new line of anticancer treatment).
  Arms: Group "Placebo"

SUMMARY:
Melatonin may represent an effective complementary treatment to standard anticancer treatments in order to reduce asthenia, depression, sleep disturbances, cognitive impairment and performance status as part of quality of life. Moreover, melatonin has been evaluated in several clinical trials in cancer patients with no side effects. It could be particularly of interest in elderly cancer patients as they exhibit a significant deficiency of melatonin production .

The investigators propose to perform a prospective and randomized study to study the effect of a melatonin supplementation on the quality of life of elderly advanced/metastatic cancer patients (age ≥ 70) treated for a locally advanced or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > = 70 years.
* Performance status < = 2 (WHO criteria)
* Life expectancy > 3months
* A patient with solid tumor locally advanced or metastatic
* Indication of systemic anticancer treatment : oral or IV chemotherapy, endocrine therapy, target therapy or immunotherapy
* MMS-orientation ≥ 7 (geriatric Mini Mental State face-to-face questionnaire)
* Able to swallow and retain oral treatment
* Patient who signed the participation consent before entering the trial
* Patient able to read, write and understand French.
* Affiliation to the french social security scheme (or beneficiary of such a scheme) under the terms of the law of 9 August 2004.

Exclusion Criteria:

* Haematological cancers
* Renal failure or hepatic failure
* Auto-immune disease
* Diagnosed neurodegenerative diseases
* Unability to fill out questionnaires
* melatonin treatment ongoing or completed for less than 3 months
* Treatment with an investigational drug, participation to another therapeutic clinical trial within <30 days
* Hypersensitivity to melatonin or any of the excipients
* Current Treatment with fluvoxamine, 5- or 8-methoxypsoralen, cimetidine, estrogen
* A history of known or suspected excessive alcohol use.
* Patient refusing to participate and / or unable to give informed consent
* Patient unable to complete the questionnaires even with the help of a relative or a nurse
* Patient does not have the capacity to comply with the study requirements
* Patient deprived of liberty by a court or administrative.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
comparison of average individual variation of overall score of QLQ-C30 of the 2 groups "Melatonin" and control (placebo) | 3 months
  The quality of life will be assessed using the QLQ-C30 questionnaire. the change in absolute value (inclusion versus after 3 months of supplementation) of overall score of QLQ-C30.

SECONDARY OUTCOMES:
Sub-scores of QLQ-C30 questionnaire especially dimensions "symptoms" and "functional" | 1 year
longitudinal evolution of QLQ-C30 scores | 1 year
Evolution of scores of QLQ-ELD14 | 1 year
sleep quality: Questionnaire Leeds | 1 year
Fatigue: visual analog scale (VAS) | 1 year
Pain: VAS | 1 year
Depression: Questionnaire GDS (Geriatric Depression Scale) | 1 year
Tolerance: assessed and graded according to the NCI-CTC (National Cancer Institute Common Toxicity Criteria) version 4.0 | 1 year
one year Overall survival rate | 1 year
one year recurrence-free survival rate | 1 year
Cognitive function: MMS (mini-mental score) or Folstein test | 1 year
Evaluation of autonomy: ADL-IADL questionnaires | 1 year
Compliance to treatment | 3 months
  counting of remaining tablets during the 3 months of supplementation
evaluation of the appetite with an EVA | 1 year
  Evaluation of the effect of melatonin on anorexia will be achieved through the evaluation of the appetite with an EVA 10 points.
evaluation of Dietary intake with dietary questionnaires | 1 year
  Dietary intake may be assessed using dietary questionnaires taken on the last 3 days, only for patients at risk of malnutrition or poor nutritional status, detected during the geriatric assessment (according to the MNA questionnaire assessing status nutritional)
Secretion of melatonin: urinary concentration of 6-sulfatoxy-melatonin (urine night 12h), with normalization on creatinuria | 3 months
Circadian rhythms of activity / rest: survey using actimeters worn for 48 hours | baseline and after 3 months of treatment
  Evaluation for only 80 patients

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, Pr, Principal Investigator — Centre Jean Perrin
Locations (12):
- France (12):
  - Institut de Cancérologie de l'ouest - Site Paul Papin, Angers
  - CHU Besançon, Besançon
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon-Bérard, Lyon
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Jean Godinot, Reims
  - Institut de Cancérologie de l'ouest - Site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Hôpital Paul-Brousse, Villejuif

REFERENCES:
- [Derived] Ginzac A, Bourbouloux E, Rivoirard R, Jouannaud C, Hager MO, Dubois S, Kwiatkowski F, Molnar I, Thivat E, Durando X. Melatonin supplementation for quality of life in older patients with advanced cancer: a randomized controlled trial. BMC Geriatr. 2025 Dec 20. doi: 10.1186/s12877-025-06899-1. Online ahead of print. PMID 41421991